CLINICAL TRIAL: NCT02201641
Title: Efficacy of Calcium Silicate Pulp-capping; a Randomized Controlled Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-LO-1893
Record Dates: First submitted 2014-07-23; First posted 2014-07-28 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Reversible Pulpitis
Keywords: Indirect pulp capping; reversible pulpitis; periapical radiolucency; periapical radiographs; cone beam computed tomography; calcium silicate cements; glass ionomer cements; caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- calcium silicate cement (Biodentine™) (Experimental): calcium silicate cement (Biodentine™) used for indirect pulp capping of teeth with deep carious lesions and inflammed pulps.
  Interventions: Device: calcium silicate cement (Biodentine™)
- Cone Beam computed tomography (CBCT) (Experimental): CBCT scans are taken to assess the efficacy of this method in detecting the presence of early peri-radicular lesions.
  Interventions: Radiation: Cone Beam computed tomography (Morita Accuitomo)
- Periapical radiographs (Active Comparator): Periapical radiographs are taken as a control to detect the presence of early peri-radicular lesions.
  Interventions: Radiation: Periapical radiographs
- Glass ionomer cement ( Fuji IX™) (Active Comparator): Glass ionomer cement ( Fuji IX™) used for indirect pulp capping of teeth with deep carious lesions and inflammed pulps.
  Interventions: Device: glass ionomer cement ( Fuji IX™)

INTERVENTIONS:
Radiation: Cone Beam computed tomography (Morita Accuitomo) — CBCT scans are taken to assess the efficacy of this method in detecting the presence of early peri-radicular lesions.
  Arms: Cone Beam computed tomography (CBCT)
Radiation: Periapical radiographs — Periapical radiographs are taken as a control to detect the presence of early peri-radicular lesions.
  Arms: Periapical radiographs
Device: calcium silicate cement (Biodentine™) — calcium silicate cement (Biodentine™) used for indirect pulp capping of teeth with deep carious lesions and inflammed pulps.
  Arms: calcium silicate cement (Biodentine™)
Device: glass ionomer cement ( Fuji IX™) — glass ionomer cement ( Fuji IX™) used for indirect pulp capping of teeth with deep carious lesions and inflammed pulp.
  Arms: Glass ionomer cement ( Fuji IX™)

SUMMARY:
This study aims to investigate the tooth nerve response to a recently introduced therapeutic filling material (calcium silicate cement) called Biodentine and to assess the quality of the overlying filling compared to another material (glass ionomer cement) called Fuji IX used more commonly. Also to compare the effectiveness of cone beam computed tomography x-rays compared to conventional periapical x-rays in detecting lesions around these teeth.

DETAILED DESCRIPTION:
Tooth decay is one of the most widespread diseases in the world. Very often, a patient comes to the dental clinic when experiencing pain which commonly means the decay is deep and is very close to or has penetrated the nerve of the tooth. When the decay is very close to the pulp or nerve of the tooth, a procedure called pulp capping is done in an attempt to save the tooth and to prevent root canal treatment. A material has been introduced to the market for this purpose, called Biodentine. This study aims to investigate the nerve response to this material and to assess the quality of the overlying filling compared to another material (glass ionomer cement) used more commonly. Also, X-rays are a routine procedure used to assess how close the decay is to the nerve and to see if there are abnormalities around the tooth. However conventional X-rays may not be accurate. A new technique called Cone Beam Computed Tomography (CBCT) has been developed which shows a 3-D image of the tooth and may be more accurate. We aim to compare the images gained from conventional X-rays and CBCT to help improve diagnosis and care planning for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients either male or female over the age of 16 (who can consent for themselves) in good general health
2. A minimum of one carious lesion (occlusal, proximal, or MOD)
3. Positive pulp response to electric pulp test and thermal stimulation.

Exclusion Criteria:

1. Patients with clinical symptoms of irreversible pulpitis who need root canal treatment
2. The presence of fistulas or swelling
3. Anterior teeth with aesthetic concerns
4. External or internal root resorption
5. Multiple teeth with carious lesions in the same quadrant,
6. Mobile teeth or tenderness to percussion.
7. Pregnant women, in view of requirements for radiographs.
8. Patients younger than 16.
9. Patients unable to give consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The principal outcome of the study is whether the tooth restored with the test or control material remains vital (alive) at follow-up examination. | up to 2 years
  The vitality of the restored tooth (whether the nerve of the tooth is alive or dead) is determined clinically by a positive response to cold test, absence of spontaneous pain, negative sensitivity to percussion, absence of sinus/fistula/swelling and abnormal mobility, and absence/reduction of periapical radiolucencies as determined by PA radiographs.

SECONDARY OUTCOMES:
The integrity of the composite restoration overlying the test or control material is either acceptable or not. | up to 2 years
  As assessed clinically by USPHS criteria and Hickel's criteria for the assessment of dental restorations.
The CBCT scans of the teeth restored with the test or control material are either more effective or are comparable to conventional radiographs in detecting the presence of early peri-radicular lesions associated with the restored teeth. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F Watson, BDS,MSc,PhD, Study Chair — King's College London
Locations (1):
- King's College Dental Institute at Guy's Hospital, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hashem D, Mannocci F, Patel S, Manoharan A, Watson TF, Banerjee A. Evaluation of the efficacy of calcium silicate vs. glass ionomer cement indirect pulp capping and restoration assessment criteria: a randomised controlled clinical trial-2-year results. Clin Oral Investig. 2019 Apr;23(4):1931-1939. doi: 10.1007/s00784-018-2638-0. Epub 2018 Sep 19. PMID 30232625
- [Derived] Hashem D, Mannocci F, Patel S, Manoharan A, Brown JE, Watson TF, Banerjee A. Clinical and radiographic assessment of the efficacy of calcium silicate indirect pulp capping: a randomized controlled clinical trial. J Dent Res. 2015 Apr;94(4):562-8. doi: 10.1177/0022034515571415. Epub 2015 Feb 20. PMID 25710953